CLINICAL TRIAL: NCT02400879
Title: Comparisons of Postoperative BIS Profile and Extubation Time After Valvular Heart Surgery: Remifentanil-based Propofol-supplemented Versus Sevoflurane-sufentanil Balanced Anesthesia Regimen
Brief Title: Remifentanil Anesthesia and Postoperative BIS in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KUH-1160080
Record Dates: First submitted 2015-03-15; First posted 2015-03-27 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Disease
Keywords: bispectral index; cardiac surgery; recovery; remifentanil
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Remifentanil; halofantrine; Sevoflurane; Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil (Active Comparator): For anesthesia maintenance, TCI-remifentanil (fixed Cp of 20 ng/ml) and TCI-propofol (variable Ce < 2.0 µg/ml) for maintaining BIS 40-60
  Interventions: Drug: Remifentanil
- sevoflurane and sufentanil (Placebo Comparator): TCI-sufentnail (Cp of 0.4-0.8 ng/ml) and sevoflurane (< 1.5 MAC) for maintaining 80-120 % of preoperative value and BIS < 60
  Interventions: Drug: sevoflurane and sufentanil

INTERVENTIONS:
Drug: Remifentanil — administering remifentanil infusion 0.7-0.8 mcg/kg/min for anesthesia maintenance
  Other Names: ultiva, GSK
  Arms: Remifentanil
Drug: sevoflurane and sufentanil — administering sevoflurane and sufentanil for anesthesia maintenance
  Other Names: sevorane and sufental
  Arms: sevoflurane and sufentanil

SUMMARY:
Background: Although remifentanil based anesthesia has been preferred for fast-track cardiac anesthesia, its recovery profile in cognitive function has not been investigated. Authors determined postoperative Bispectral index (BIS) score as well as extubation time after remifentanil-based propofol-supplemented anesthesia and compared them with those after conventional balanced sevoflurane-sufentanil anesthesia.

Methods: Patients undergoing cardiac surgery using moderate hypothermic cardiopulmonary bypass (CPB) will be randomly allocated to get remifentanil-based propofol-supplemented (Group R) or conventional sevoflurane-sufentanil regimen (Group C) in the study period. For anesthetic induction and maintenance, fixed target controlled infusion (TCI) of remifentanil (plasma concentration 20 ng/ml) and TCI-propofol for maintaining BIS score 40-60 (effect concentration 0.8-1.5 μg/ml) in Group R, and TCI-sufentanil (Cp 0.4- 0.8 ng/ml) and sevoflurane inhalation for maintaining 80-120 % of baseline BP and BIS < 60 (< 1.5 MAC) in Group C, respectively.

Authors will analyze postoperative recovery of cognitive function by using BIS after the use of remifentanil-based propofol-supplemented anesthesia for cardiac surgery and to compare them to those after the use of conventional balanced sevoflurane-sufentanil anesthesia.

DETAILED DESCRIPTION:
Backgrounds Since opioid-based anesthesia does not produce dose-dependent myocardial depression, it has been applied for patients undergoing cardiac surgery with myocardial dysfunction.

However, prolonged use of conventional opioids in a large dosage delays patient's postoperative recovery due to their longer half-life and accumulation of their metabolites.

Fast-track cardiac anesthesia which reducing the duration of postoperative mechanical ventilation and length of stay (LOS) in the intensive care unit (ICU) is beneficial not only in reducing ventilator-related complications and medical expense but in improving patient's outcome.

For this purpose, in addition to supplementation of neuraxial blockade, use of short-acing opioid, such as remifentanil, has been advocated for cardiac anesthesia. Remifentanil is an ultra-short acting opioid and provides not only stable hemodynamics, as other opioid does, and but fast recovery, even after prolonged use in a large dosage. In further, recent investigations showed that remifentanil provides preconditioning effect in myocardial ischemia injury during cardiac surgery, as like in the use of volatile anesthetics including sevoflurane.

Remifentanil vs volatile anesthetics In spite of the importance of recovery of cognitive function on whole postoperative clinical features, most investigations have evaluated only the postoperative respiratory profile in determining the speed of postoperative recovery specific to the choice of anesthesia regimen.

Bispectral index (BIS) monitoring has been used to monitor sedation depth, to avoid introperative awareness and to adjust the dosage of intraoperative hypnotics. Several investigations tried to find BIS's efficacy in managing sedation of critically ill patients. In spite of some controversies, BIS monitoring seem to be beneficial: it does not require additional stimuli to determine sedation level which is essential in other subjective modalities, such as Ramsay score, and usually compromises the already instituted patient's sedation level.

Authors will analyze postoperative recovery of cognitive function by using BIS as well as respiratory profiles after the use of remifentanil-based propofol-supplemented anesthesia for cardiac surgery and to compare them to those after the use of conventional balanced sevoflurane-sufentanil anesthesia.

Methods Population and Study Protocol After obtaining Institutional Review Board approval and informed consents from the patients, they are prospectively studied among patients undergoing cardiac valve repair or replacement surgery under moderate hypothermic cardiopulmonary bypass (CPB).

During the study period (6 months), at least, forty patients are randomly allocated into following one of two groups using sealed envelopes: remifentanil-based propofol-supplemented anesthesia regimen is employed in Group R and conventional balanced sevoflurane-sufentanil anesthesia regimen in Group C, respectively.

Preoperative and intraoperative exclusion criteria Preoperative exclusion criteria 1) urgent or emergent surgery, 2) left ventricle (LV) ejection fraction < 50%, 3) application of intraaortic balloon pump (IABP), 4) myocardial infarction, 5) neurologic deficit, 6) hepatic or renal impairment, 7) pacing, 8) inotropic medication, 9) neurologic deficit.

Intraoperative exclusion criteria

1) CPB application > 250 min, 2) transfused of packed red blood cell (pRBC) > 5 units, 3) post-CPB use of double inotropic support > 30 min , 4) post-CPB pacing, 5) IABP 6) IABP 7) postoperative hemodialysis, 8) excessive bleeding > 750 ml during postoperative 6 hour, 9) reoperation due to excessive bleeding.

All data were collected by trained observers who did not participate in patient care and who were blinded to the current study.

Anesthesia regimen After establishing routine invasive arterial blood pressure and noninvasive patient monitoring such as pulse oximetry (SpO2), electrocardiography, bispectral index (BIS) and cerebral oximetry, anesthesia is induced by two staff anesthesiologist (AA and BB) using a target controlled infusion (TCI) of propofol (effect site concentration, Ce, of 2.0 µg/ml) and remifentanil (plasma concentration, Cp, of 20 ng/ml with the time to reach target concentration of 7 min) in Group R (by AA), and anesthesia is induced by bolus injection of thiopental sodium 3-4 mg/kg and maintained using TCI- sufentanil (Cp of 0.4 ng/ml) in Group C (by BB). Muscle relaxation and tracheal intubation is facilitated by bolus rocuronium under the guidance of peripheral neuromuscular transmission.

For anesthesia maintenance, TCI-remifentanil (fixed Cp of 20 ng/ml) and TCI-propofol (variable Ce < 2.0 µg/ml) for maintaining BIS 40-60 in Group R [14], and TCI-sufentnail (Cp of 0.4-0.8 ng/ml) and sevoflurane (< 1.5 MAC) for maintaining 80-120 % of preoperative value and BIS < 60 in Group C, respectively. Rocuronium is continuously infused (3 µg/kg/min) in both groups.

Controlled ventilation of O2/air mixture (FiO2 0.5-0.6) is performed with following setting of anesthesia ventilator (ADU™, Datex-Ohmeda, Finland): tidal volume of 7 ml/ideal body weight (calculated by obsolete formulas), respiratory rate maintain normocarbia (end-tidal CO2 tension 35-40 mmHg) and inspiratory:expiratory ratio of 1:2.

Pulmonary artery catheter (Swan-GanzCCOmboCCO/SvO2, Edwards Lifesciences, Irvine, USA) and a probe of transesophageal echocardiography were placed after anesthesia induction.

If high BIS score (> 60) persisted against the increase of sevoflurane to 1.5 MAC in Group C or Ce of propofol to 2.0 μg/ml in Group R, bolus midazolam 2 mg is administered.

Surgery and CPB regimen All surgery is performed by one surgeon and 4 surgical assistants. After performing sternotomy and administration of heparin 300 units/kg, arterial and venous cannulations for CPB are performed at activated clotting time (ACT) > 450 sec and CPB was conducted using reservoir, membrane oxygenator, roller pump and heat exchanger. Priming volume for CPB was composed of normal saline, 20% mannitol, NaHCO3, 20% albumin, heparin, antibiotics and calcium gluconate. The flow of CPB is initiated at 60 ml/kg/min and adjusted by the current hemodilution and temperature.

Antegrade or retrograde administration of cold cardioplegic solution (20 ml/kg) consisting of drained patient's blood, NaCl 6.43 g/L, KCl 1.193 g/L, CaCl2 0.176 g/L and MgCl2 3.253 g/L (pH 7.4 at 4 - 8 °C) is applied as appropriate for cardiac protection after application of aortic cross clamp (ACC).

Transfer to intensive care unit (ICU) and postoperative pain control After surgery, the patients are transferred to the ICU in intubated status and received controlled or assisted ventilation till the time of extubation. In Group R, remifentanil 0.25-0.3 μg /kg/min is continued till the time of extubation.

For postoperative pain control, the intravenous patient control analgesia consisting of alfentanil, ketorolac, and ondansetron is started at the time of sterna closure in Group C or at 20 min before extubation in Group R, respectively.

Protocols of ventilator weaning and extubation The mode of ventilator is converted from volume controled ventilation (CMV) to synchronized intermittent mandatory ventilation (SIMV) when the following criteria were achieved: stable hemodynamics, self respiration, and the respiratory rate 10-25 breaths/min [15].

The patients are extubated when the following criteria are achieved: awake state, stable hemodynamics, normal airway reflex, respiratory rate 10-25 breath/min, SpO2 > 95% at FiO2 < 0.6, pH ≥ 7.3 and PaCO2 < 55 mmHg.

Measurements Operation time, CPB time, ACC time, intraoperative fluid administration quantity, transfusion requirements, intraoperative urine output (UO), preoperative and postoperative hematocrit (Hct) and preoperative and postoperative PaO2/FiO2 ratio are recorded.

The duration from the end of surgery to the time of achieving BIS score > 80 (persisting > 3 min) (T-BIS80) [16], the duration from end of surgery to the time of initiating SIMV (T-SIMV) and the duration from the end of surgery to the time of extubation (T-extubation) are measured.

Statistical analysis The primary outcome variables are T-BIS80, T-SIMV, and T-extubation. Statistics are performed using the program Sigmastat ver.3.1(Systat Software Inc, San Jose, USA). Continuous variables were analyzed by a t-test, while categorical variables are by a chi-square test between two groups. The data collected are expressed as mean and standard deviation, numbers of patients or absolute numbers. A P value < 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing cardiac valve repair or replacement surgery under moderate hypothermic cardiopulmonary bypass (CPB).
2. All patients should provide written informed consents

Exclusion Criteria:

Preoperative exclusion criteria

1. urgent or emergent surgery,
2. left ventricle (LV) ejection fraction < 50%,
3. application of intraaortic balloon pump (IABP),
4. myocardial infarction,
5. neurologic deficit,
6. hepatic or renal impairment,
7. pacing,
8. inotropic medication,
9. neurologic deficit.

Intraoperative exclusion criteria

1. CPB application > 250 min,
2. transfused of packed red blood cell (pRBC) > 5 units,
3. post-CPB use of double inotropic support > 30 min ,
4. post-CPB pacing,
5. IABP
6. IABP
7. postoperative hemodialysis,
8. excessive bleeding > 750 ml during postoperative 6 hour,
9. reoperation due to excessive bleeding.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
time to achieving BIS>80 | 5 min
  The duration from the end of surgery to the time of achieving BIS score > 80 (BIS>80 persisting > 3 min)

SECONDARY OUTCOMES:
time to achieve SIMV ventilation mode | 5 min
  the duration from end of surgery to the time of initiating SIMV (T-SIMV)
time to achieve extubation | 5 min
  the duration from the end of surgery to the time of extubation (T-extubation)

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk Univeristy Medical Center